CLINICAL TRIAL: NCT04424524
Title: An Implementation Project to Improve the Efficiency of PrEP Delivery in Public Health HIV Care Clinics in Kenya
Brief Title: Streamlining the Efficiency of PrEP Implementation
Acronym: Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kenneth K Mugwanya, Assistant Professor, School of Medicine: Global Health, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00007949; R00MH118134 (NIH)
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: HIV Prevention; HIV Preexposure Prophylaxis; Implementation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct-to-pharmacy oral PrEP refill visits (Other): Intervention
  Interventions: Other: Direct-to-pharmacy oral PrEP refill visits
- Usual care (No Intervention): Control

INTERVENTIONS:
Other: Direct-to-pharmacy oral PrEP refill visits — Programmatic direct-to-pharmacy oral PrEP refill visits supported with client HIV self-testing
  Arms: Direct-to-pharmacy oral PrEP refill visits

SUMMARY:
This is a pilot facility-based direct-to-pharmacy PrEP refill delivery to streamline care pathway in Kenyan public health HIV facilities implementing PrEP. Data on up to 500 PrEP users will be evaluated to understand delivery efficiency and in-depth interview with users and delivery key informants will be conducted to identify barriers and facilitators of implementation.

DETAILED DESCRIPTION:
A prospective, pilot implementation evaluation of patient-centered differentiated care service. The core components of the multifaceted implementation strategy include: 1) 3-monthly refills, 2) direct-to-pharmacy refill visits, 3) HIV self-testing (HIVST) while waiting for refills, 4) Rapid risk assessment for ongoing risk, adherence, side effect, and acute HIV symptoms. Clinics will implement either: 1) current PrEP patient flow without any change or 2) a pilot differentiated pharmacy-based follow up PrEP care pathway. Clinics will implement only one delivery model thus eliminating risk for confusion in the clinic about delivery models and permitting a full-scale test of the system, since the efficiency in PrEP delivery is in part at the system level, above and beyond the individual client encounter. For this pilot project designed to primarily test delivery efficiency, feasibility and acceptability of direct-to-pharmacy care pathway at systems level using existing public health infrastructure, pilot and control clinics will be of comparable size selected to reflect the implementation nature of the design.

The specific aims are:

Aim 1: To evaluate whether a differentiated care model improves the efficiency of PrEP delivery while resulting in equivalent or better: 1) patient waiting time, 2) early PrEP continuation, and 3) adherence.

Aim 2: Conduct mixed-methods study to understand patient and provider perception, experiences , feasibility and acceptability of a differentiated PrEP delivery model.

Aim 3: Assess the efficiency, cost and cost-effectiveness of a facility-based differentiated PrEP care.

ELIGIBILITY:
Inclusion Criteria:

For HIV-negative participants:

* Of legal age (≥18 years)
* Able and willing to provide written informed consent for research component of the project (blood draw for adherence, brief surveys and in-depth qualitative interviews)
* HIV uninfected based on negative HIV tests, per Kenya national guidelines
* Currently or previously accessed PrEP at participating HIV clinic

For Key delivery informants:

* Able willing and able to provide consent in order to participate in the survey and qualitative interviews.
* Works at any of the clinics implementing PrEP delivery. Key informants may include HIV testing service nurses, counselors, clinicians, social workers, or clinic managers.

Exclusion Criteria:

* Not meeting any of the inclusion criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Patient wait time | up to 6 months
  Total waiting time at the clinic and contact time with providers measured by time and motion studies
PrEP continuation | up to 6 months
  Measured by return to clinic for PrEP refill
PrEP adherence | up to 6 months
  Measured objectively through tenofovir levels in dried blood spots at random subset of PrEP visits
Acceptability of direct-to-pharmacy PrEP care pathway | up to 6 months
  Assessed by the Acceptability of Intervention Psychometric Measure (AIM)
Acceptability of user HIV self-testing for PrEP care pathway | up to 6 months
  Assessed by the Acceptability of Intervention Psychometric Measure (AIM)
Feasibility of direct-to-pharmacy PrEP care pathway | up to 6 months
  Assessed by the Feasibility of Intervention Psychometric Measure (FIM)

SECONDARY OUTCOMES:
Barriers to implementation of direct-to-pharmacy PrEP care pathway in Kenyan public health HIV clinics | up to 6 months
  Evaluated through in-depth and key informants qualitative interviews
Facilitators to implementation of direct-to-pharmacy PrEP care pathway in Kenyan public health HIV clinics | up to 6 months
  Evaluated through in-depth and key informants qualitative interviews
Fidelity of implementing of direct-to-pharmacy PrEP care pathway in Kenyan public health HIV clinics | up to 6 months
  Extent to which core components of the direct-to-pharmacy PrEP care pathway are implemented as intended will be evaluated through checklists and surveys with clinic managers
Safety of HIV self-testing | up to 6 moths
  Accuracy of HIV self-testing measured by frequency false negative and positive tests.
Reasons for PrEP discontinuation | up to 6 months
  Measured through in-depth qualitative interviews and surveys with persons who discontinue PrEP use
Cost of implementing direct-to-pharmacy PrEP care pathway in Kenyan public health HIV clinics | up to 6 months
  Measured through micro-activity costing and time and motion studies

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Mugwanya, MBChB, PhD, Principal Investigator — University of Washington
Locations (1):
- Partners in Health Research and Development, Thika, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Data from Streamlining Efficiency of PrEP Implementation Study will be available by contacting the International Clinical Research Center at the University of Washington (icrc@uw.edu)
Time Frame: After primary results are reported

REFERENCES:
- [Result] Zewdie KB, Ngure K, Mwangi M, Mwangi D, Maina S, Etyang L, Maina G, Ogello V, Owidi E, Mugo NR, Baeten JM, Mugwanya KK. Effect of differentiated direct-to-pharmacy PrEP refill visits supported with client HIV self-testing on clinic visit time and early PrEP continuation. J Int AIDS Soc. 2024 Mar;27(3):e26222. doi: 10.1002/jia2.26222. PMID 38446643
- [Derived] Wairimu N, Ngure K, Ogello V, Owidi E, Mwangi P, Etyang L, Waituika W, Mwangi M, Githuku DM, Maina S, Irungu E, Mugo N, Mugwanya KK. Low HIV-risk aligned discontinuation among HIV pre-exposure prophylaxis users within public HIV clinics in Kenya: A mixed method study. PLOS Glob Public Health. 2025 Apr 28;5(4):e0004493. doi: 10.1371/journal.pgph.0004493. eCollection 2025. PMID 40294082